CLINICAL TRIAL: NCT06938425
Title: Effectiveness of Intratissue Percutaneous Electrolysis and Deep Dry Needling Versus a Standard Physical Therapy Protocol in the Treatment of Whiplash Syndrome in the Short and Medium Term
Brief Title: Effectiveness of Percutaneous Electrolysis and Dry Needling vs. Standard Therapy for Whiplash Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Camilo Jose Cela University (Other)
Responsible Party: Principal Investigator, Rocío Fernández Navarro, Principal investigator, Camilo Jose Cela University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 16_23_FINER
Record Dates: First submitted 2025-02-03; First posted 2025-04-22 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Whiplash Injuries
Keywords: Percutaneous electrolysis; Dry needling; Whiplash; Myofascial pain syndrome; Myofascial trigger point; Intrafibrillar blood flow; elasticity
MeSH Terms: conditions — Whiplash Injuries; Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- standard physiotherapy treatment (Active Comparator): Participants in this group will receive standard physical therapy sessions, including manual techniques, massage therapy and mobility exercises.
  Interventions: Procedure: Standard physiotherapy
- intratissue percutaneous electrolysis (Experimental): Participants in this group will receive physiotherapy sessions using the Percutaneous Intratisular Electrolysis (EPI) technique,
  Interventions: Other: intratissue percutaneous electrolysis
- Deep Dry needling (Experimental): Participants in this group will receive physiotherapy sessions using the dry puncture technique applied to active trigger points.
  Interventions: Other: deep dry needling

INTERVENTIONS:
Other: intratissue percutaneous electrolysis — Using fine needles guided by ultrasound to apply electrical stimulation directly to the affected tissue (for example, damaged muscles or tendons).
  Arms: intratissue percutaneous electrolysis
Other: deep dry needling — Insertion of fine needles into muscle trigger points (without injection of drugs) to relieve muscle pain and release tension.
  Arms: Deep Dry needling
Procedure: Standard physiotherapy — It includes manual techniques such as therapeutic massage and mobilization, along with stretching and strengthening exercises to improve range of motion and reduce pain.
  Arms: standard physiotherapy treatment

SUMMARY:
The main objective of this research is to evaluate the effectiveness of two interventions (PIE vs DDN) in adult patients who have suffered a LCS after a traffic accident and comparing it with a standard physiotherapy program. As a secondary objective, the investigators will analyze the reduction of intrafibrillar blood flow and muscle elasticity perceived by the patient in the long term and the reduction of pain and disability appreciated by the patient.

It is hypothesized as an alternative hypothesis that percutaneous electrolysis and/or deep dry needling intervention in combination with standard physiotherapy will give better clinical outcomes in patients with active trigger point LCS following a road traffic accident compared to the current standard physiotherapy intervention.

The researchers will compare both invasive physical therapy techniques with standard treatment to see if these techniques are more effective in treating whiplash syndrome.

DETAILED DESCRIPTION:
The present study primarily aims to evaluate the clinical effectiveness of two invasive physiotherapy techniques-percutaneous intratissue electrolysis (PIE) and deep dry needling (DDN)-combined with conventional physiotherapy, compared to a standard physiotherapy program in adult patients who have sustained a whiplash-associated disorder (WAD) following a motor vehicle accident.

Whiplash injury is one of the most common musculoskeletal sequelae after traffic accidents, often leading to chronic pain and functional disability. The heterogeneity of clinical responses and the persistence of symptoms underscore the need for optimized therapeutic strategies supported by high-quality evidence.

This prospective, randomized controlled trial (RCT) will include three parallel intervention arms:

Control group: standard physiotherapy based on therapeutic exercise and manual therapy techniques.

Experimental group 1: standard physiotherapy + PIE intervention.

Experimental group 2: standard physiotherapy + DDN intervention.

The study population will consist of adult subjects diagnosed with WAD and the presence of active myofascial trigger points in the cervical musculature. Participants will be randomly assigned to one of the three groups, and interventions will be administered over a predetermined period, with follow-up assessments scheduled at both short- and long-term intervals.

Secondary outcomes include:

Changes in intrafibrillar blood flow Patient-reported muscle elasticity, Self-reported pain levels Functional disability

The alternative hypothesis proposes that the application of invasive techniques (PIE or DDN) as an adjunct to conventional physiotherapy will yield superior clinical outcomes in terms of pain reduction, functional improvement, and muscle parameter normalization when compared to standard physiotherapy alone.

This study aims to generate robust scientific evidence regarding the comparative efficacy of these interventions and to inform clinical decision-making in the rehabilitative management of post-traumatic whiplash-associated disorders.

ELIGIBILITY:
Inclusion Criteria:

* Adults with whiplash syndrome following a traffic accident.
* Patients must reside or stay in the Autonomous Community of Melilla during the intervention phase.
* Subjects will have the presence of neck pain after suffering a traffic accident and the presence of at least one active trigger point in the sternocleidomastoid and/or levator scapulae muscles.
* All subjects who suffer a traffic accident and who have a score of 5 or higher on the numerical scale (EN) of pain assessment.

Exclusion Criteria:

* Patients undergoing anticoagulant treatment.
* Patients who have suffered previous cervical trauma or who have undergone surgery in the last year.
* Subjects who present some type of alteration (skin or infection, sensitivity or pain perception).
* Subjects with central or peripheral nervous system involvement.
* Patients who have problems with the material: allergy to metal, belonephobia (fear of needles).
* Pregnant women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Intrafibrillar blood flow | From the beginning of treatment to the end of treatment at 4 weeks and at 3 months
  To assess intrafibrillar blood flow, the ultrasound tool is used, with color Doppler. the hypervascularity of small vessels in the inflamed synovial tissue of the structures is evaluated. Measurements are expressed in liters per minute (l/min).
Elasticity of muscle fibers | From the beginning of treatment to the end of treatment at 4 weeks and at 3 months
  Elastography is used to evaluate the elasticity of muscle fibers. It is a grayscale ultrasound technique that is superimposed on the color parametric image that expresses the rate of tissue deformation.Making it possible to express the stiffness and elasticity of the tissue in units of pressure (kilopascals).

SECONDARY OUTCOMES:
Pain perceived by the patient | From the beginning of treatment to the end of treatment at 4 weeks and at 3 months
  Pain is a quantitative variable. The investigators will use the numerical evaluation scale (EN), which consists of a numbered scale from 1 -10.
Pain perceived by the patient | From the beginning of treatment to the end of treatment at 4 weeks and at 3 months
  Another pain variable is the pressure pain threshold (PPT), which is an unpleasant sensory and emotional experience associated with a present injury and a pressure algometer will be used. Measurements are expressed in kg/cm2.
Disability | From the beginning of treatment to the end of treatment at 4 weeks and at 3 months
  To assess disability, the investigators will use the Whiplash Disability Questionnaire (WDQ) scale. It is the first instrument for patients with whiplash syndrome, which includes items related to areas of life, personal care and work and those related to the perception of pain. This questionnaire consists of 13 items, scored from 0 to 10 points.

CONTACTS AND LOCATIONS:
Overall Officials: María Benito, PhD, Study Director — Associate Professor

REFERENCES:
- [Derived] Fernandez-Navarro R, Benito-de-Pedro M, Navarro Reyes FM, Moreno-Lopez J, Estebanez-Perez MJ, Pastora-Bernal JM. Intratissue percutaneous electrolysis and deep dry needling compared to a standard physiotherapy protocol in the treatment of whiplash syndrome: study protocol for a randomized controlled trial. Front Rehabil Sci. 2025 Nov 3;6:1670603. doi: 10.3389/fresc.2025.1670603. eCollection 2025. PMID 41255411